CLINICAL TRIAL: NCT02997527
Title: Measurement of the Distal 5 cm of the Esophagus in Patients With Non-Erosive Reflux Disease and Controls
Brief Title: [Impedance Measurement for Non-Erosive Reflux Disease
Acronym: Impedance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Completed very similar study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, David A. Kazka, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-007762
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: GERD; Healthy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Acoustic Impedance Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraluminal impedance testing (Experimental): During the participant's clinical endoscopy the 2.13 mm catheter (tiny tube), called an Intraluminal Impedance, will be passed through the channel of the standard endoscope.
  * The catheter (tiny tube) will be placed through the endoscope in your esophagus 1 cm above where your stomach and esophagus meet for 5 seconds.
  * At 2 cm above where your stomach and esophagus meet the catheter will be placed for 5 seconds
  * And at 3 cm above where the participants stomach and esophagus meet the catheter will be placed for 5 seconds.
  * At 4 cm above where the participants stomach and esophagus meet the catheter will be placed for 5 seconds.
  * At 5 cm above where the participants stomach and esophagus meet the catheter will be placed for 5 seconds.
  Interventions: Device: Intraluminal Impedance

INTERVENTIONS:
Device: Intraluminal Impedance — Esophageal impedance testing measures epithelial integrity as reflected through the ability of the mucosa to conduct electric current. Recently, a site specific endoscopically placed impedance probe has been developed that can measure esophageal mucosal impedance at any point of the esophagus.
  Other Names: Impedance testing

SUMMARY:
This study is being done to determine if people with and without GERD or trouble swallowing have increased esophageal mucosa impedance (food getting into the esophageal tissue).

DETAILED DESCRIPTION:
In patients with gastroesophageal reflux disease (GERD) but without gross evidence of esophageal injury, confirmation of acid reflux is typically performed through testing that measures reflux at or proximal to 5 cm above the gastroesophageal junction. These tests such as pH/impedance monitoring and Bravo probe placement in the esophagus have been the gold standard for diagnosing and quantitating the degree of gastroesophageal reflux. This stands in contrast to the concept that the esophagus distal to 5 cm is first and foremost exposed to gastroesophageal reflux and that most injury in the form of erosive esophagitis is seen in the 4cm segment below where this instruments measure reflux. As a result, this type of testing may not allow for full understanding of the pathophysiology of GERD. Furthermore, with refluxed acid exposure limited to the distal esophagus in some patients, use of conventional pH testing could lead to inaccurate diagnosing of GERD.

Esophageal impedance testing measures epithelial integrity as reflected through the ability of the mucosa to conduct electric current. As dilation of intercellular spaces in biopsies from patients with GERD is considered the earliest indication of esophageal injury in response to reflux in the absence of gross endoscopic injury, the measure of increased current conduction through these dilated spaces has been shown to be an accurate means of diagnosing patients with non-erosive reflux disease. To this point, most esophageal impedance has been measured using impedance ports placed at locations similar to the pH probes in a combined intra-esophageal ambulatory catheter. As a result, the most distal point of impedance measurement is also 5 cm above the gastroesophageal junction. Recently, a site specific endoscopically placed impedance probe has been developed that can measure esophageal mucosal impedance at any point of the esophagus.

In this study the Principal Investigator would like to look at patients with and without reflux symptoms measuring impedance at 1,2,3,4 and 5 cm at the 6 o'clock position above the Gastroesophageal Junction.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-90
* Patients with heartburn and no hiatal hernia undergoing clinically indicated endoscopy
* Patients with heartburn and a hiatal hernia > 3cm undergoing clinically indicated endoscopy
* Patients undergoing clinically indicated upper endoscopy for indications other than dysphagia or GERD
* Patients with reflux symptoms, a normal appearing esophagus on clinically indicated endoscopy undergoing clinically indicated ambulatory pH/impedance testing.

Exclusion Criteria:

* Previous gastric or esophageal surgery.
* Use of proton pump inhibitors 1 month prior to the study
* Patients on anticoagulation other than aspirin or clopidogrel
* Presence of erosive esophagitis or Barrett's esophagus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Epithelial integrity in GERD an Non-GERD subjects | 1 year
  A special sensor array (Mucosal Impedance) composed of 360_ circumferential sensing rings was engineered and mounted on a 2-mm-diameter soft catheter easily traversable through the working channel of an upper endoscope. The frequency for the measuring circuit was set at 2 kHz. Impedance measurements of the esophageal mucosa were expressed in ohms as the ratio of voltage to the current, according to Ohm's law (voltage ¼ IR). Data will be acquired with a stationary impedance data acquisition system and viewed and analyzed on BioView Analysis software. Impedance measurements will be obtained at 1,2,3,4, 5 cm at the 6 O'clock position above the gastroesophageal junction

SECONDARY OUTCOMES:
Epithelial integrity by Mucosal Impedance verses gold standard Ambulatory pH monitoring | 1 year
  To compare the findings of esophageal impedance probe measurement to those of traditional pH monitoring in patients with NERD undergoing clinically indicated pH/impedance monitoring to determine the accuracy of the impedance probe relative to the gold standard catheter based evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: David A Katzka, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No